CLINICAL TRIAL: NCT03201549
Title: The Effects of Increased Fructose Ingestion on FGF-21 Levels in Humans
Acronym: E228
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Jody Dushay, Assistant Professor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2017P000053
Record Dates: First submitted 2017-06-27; First posted 2017-06-28 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Fasting
MeSH Terms: conditions — Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- healthy (Experimental): healthy volunteers will ingest fructose and have FGF21 levels measured
  Interventions: Dietary Supplement: oral fructose challenge

INTERVENTIONS:
Dietary Supplement: oral fructose challenge — Participants will consume fructose for two weeks and fast for 8 hours before study visits where they will drink a fructose beverage.

SUMMARY:
The primary aim of this study is to examine the effect of fructose ingestion on serum FGF-21 levels in humans.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-60
* BMI 19-25 kg/m2; 19-23 for Asian subjects
* Stable weight (variation < 3 kg within 6 months of screening visit)
* Ability to give informed consent in English
* Use of medically approved form of contraception

Exclusion Criteria:

* Fasting blood glucose >100
* Hemoglobin A1C% > 6.5%
* Fasting triglycerides >150
* Type 1 or type 2 diabetes mellitus diagnosed according to American Diabetes Association criteria
* Coronary heart disease (history of myocardial infarction, unstable angina pectoris, or congestive heart failure)
* Uncontrolled hypertension (BP > 160/100 mmHg on or off antihypertensive medication) intravenous drug use
* Recent weight loss (> 3 kg within 6 months of the screening visit)
* Gastroparesis
* Inflammatory or irritable bowel disease
* Malignancy treated with chemotherapy within the past 3 years
* Depression or psychosis requiring hospitalization
* Renal insufficiency (creatinine clearance < 40 ml/min)
* Transaminases > 2x above the normal range
* Known liver disease
* Pregnancy within 6 months of the screening visit
* Lactation
* Failure to use medically approved contraceptive methods
* History of surgery for the treatment of obesity (gastric banding, gastric bypass, gastric stapling)
* Change in dose of thyroid hormone or antithyroidal medication within 3 months of screening visit
* History of alcohol abuse within the past 5 years
* Fructose intolerance

Exclusionary medications:

* Oral steroids
* Metformin
* Weight loss medications including nonprescription supplements

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-07-30 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Change in serum FGF21 levels | 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No